CLINICAL TRIAL: NCT02017860
Title: An Open Label, Multi-center Everolimus Roll-over Protocol for Patients Who Have Completed a Previous Novartis-sponsored Everolimus Study and Are Judged by the Investigator to Benefit From Continued Everolimus Treatment.
Brief Title: Study to Collect and Assess Long-term Safety of Everolimus in Patients Who Are on Everolimus Treatment in a Novartis-sponsored Study and Are Benefiting From the Treatment as Judged by the Investigator.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRAD001C1X01B
Record Dates: First submitted 2013-12-17; First posted 2013-12-23 (Estimated); Results first posted 2020-04-30 (Actual); Last update posted 2020-04-30 (Actual); Status verified 2020-04

CONDITIONS: Neoplasms
Keywords: RAD001, everolimus, roll-over
MeSH Terms: conditions — Neoplasms | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Everolimus (Experimental): Patients who received everolimus in a Novartis-sponsored, Oncology Clinical Development & Medical Affairs (CD&MA) study that had reached its study objectives, were not progressing on the current study treatment as defined by the parent protocol and were unable to access everolimus treatment outside of a clinical trial were enrolled.
  Interventions: Drug: Everolimus

INTERVENTIONS:
Drug: Everolimus — Everolimus was provided by the investigator in 2.5 mg or 5 mg tablets for daily oral administration.

SUMMARY:
The purpose of this study was to collect and assess long-term safety of everolimus in patients who were currently receiving everolimus treatment in a Novartis-sponsored, Oncology CD&MA study that had reached its study objectives, were not progressing on the current study treatment as defined by the parent protocol, and were unable to access everolimus treatment outside of a clinical study. Parent studies eligible to participate in the roll-over study were decided by Novartis. Investigator initiated trials (IITs) were not included. The primary objective of the parent study must have been reached and the parent study must have been in the process of being completed and reported.

DETAILED DESCRIPTION:
This was a multi-center, open label study to collect and assess long-term safety of everolimus in patients being treated in current Novartis-sponsored studies and who were benefiting from treatment with everolimus judged by the investigator.There was no screening period for this study. Eligible patients were consented and started their treatment with everolimus as soon as they entered the study. Patients had to return to the study center on a yearly basis (± 3 months), but for resupply of study medication, the frequency of the receipt and dispensing followed local practice (e.g., every 2 to 3 months). The dose of everolimus was based on the investigator's judgment.

Adverse events (AEs) were collected continuously throughout the study. For the safe and effective use of everolimus, patient could return to the clinic at any given time following local practice. When AEs were observed, additional visits were arranged by investigator's discretion.

Patients continued to be treated until they were no longer benefiting from everolimus as defined in the parent protocol (disease progression), developed unacceptable toxicities, withdrew consent, were non-compliant to the protocol, the investigator felt it is no longer in the patient's best interest to continue everolimus therapy or the patient died, whichever came first.

A patient reached the end of study when everolimus treatment was permanently discontinued and the end of treatment visit had been performed. All patients were followed for AEs for 30 days after the last dose of everolimus.

The study remained open for approximately 5 years; until such time that enrolled patients no longer needed treatment with everolimus, whichever came first.

ELIGIBILITY:
Inclusion Criteria:

* Patient is currently enrolled in a Novartis-sponsored, CD&MA study receiving everolimus or everolimus plus Sandostatin LAR Depot and has fulfilled all their requirements in the parent study
* Patient is currently benefiting from treatment with everolimus, as determined by the guidelines of the parent protocol.

Exclusion Criteria:

* Patient has been permanently discontinued from everolimus study treatment in the parent study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2014-01-16 (Actual); Primary Completion 2019-04-25 (Actual); Study Completion 2019-04-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (4):
- Japan (4):
  - Novartis Investigative Site, Matsuyama, Ehime
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Osaka, Osaka
  - Novartis Investigative Site, Kitaadachi-gun, Saitama

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 4 subjects were enrolled in the study and received at least one dose of everolimus. Of the 4 subjects, 2 subjects terminated treatment due to study closure by sponsor as approximately 5 years had elapsed since first patient first visit (FPFV). One subject terminated treatment due to an Adverse Event (AE) and one subject withdrew consent.
Period: Overall Study
Arm/Group | Everolimus
Started | 4
Completed | 2
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: All 4 subjects were included in both the Full Analysis Set and Safety Set.
Arm/Group | Everolimus
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Pariticipants With Adverse Events as a Measure of Safety and Tolerability
Description: Any sign or symptom that occurs during the study treatment plus the 30 days post treatment.
Time Frame: Adverse events were collected from first dose of study treatment until end of study treatment plus 30 days post treatment, up to maximum duration of approximately 5 years.
Population: Safety Set-included all subjects who received at least one dose (partial or complete) of everolimus, and had at least one valid post-baseline safety assessment. The statement that a subject had no AEs (on the AEs eCRF) constituted a valid safety assessment.
Measure: Number; unit: Count of Participants
Arm/Group | Everolimus
Number analyzed (Participants) | 4
Count of Participants
  Participants who had at least one Adverse Event | 4
  Participants with Grade 3/4 Adverse Event | 2

ADVERSE EVENTS:
Time Frame: Adverse events were collected from first dose of study treatment until end of study treatment plus 30 days post treatment, up to maximum duration of approximately 5 years.
Description: Any sign or symptom that occurs during the study treatment plus the 30 days post treatment.
Arm/Group | Everolimus
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 1/4
Other Adverse Events (participants affected / at risk) | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Everolimus (N=4)
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Everolimus (N=4)
Pericardial effusion (Cardiac disorders) | 2
Dental caries (Gastrointestinal disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 2
Oedema peripheral (General disorders) | 2
Conjunctivitis (Infections and infestations) | 1
Dermatophytosis of nail (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 1
Rhinitis (Infections and infestations) | 2
Blood creatinine increased (Investigations) | 2
Blood phosphorus decreased (Investigations) | 1
Haemoglobin decreased (Investigations) | 1
Weight decreased (Investigations) | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 2
Aphasia (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Neuropathy peripheral (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 2
Nail disorder (Skin and subcutaneous tissue disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Statistical Analysis Plan (2015-04-20): https://cdn.clinicaltrials.gov/large-docs/60/NCT02017860/SAP_000.pdf
  • Study Protocol (2016-08-30): https://cdn.clinicaltrials.gov/large-docs/60/NCT02017860/Prot_001.pdf